CLINICAL TRIAL: NCT05921461
Title: The Use of Hemodynamic Occlusive and Vascular Response (HOVR) Technology for the Measurement of Absorption of Light in Order to Derive Changes of Perfusion and Oxygen Levels in the Foot.
Brief Title: The Use of HOVR Technology for Assessment of Blood Associated Parameters
Status: Completed | Type: Observational
Sponsor: Votis Subdermal Imaging Technologies LTD (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: PedCheck-V1-2.1
Record Dates: First submitted 2023-05-10; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control NON-PAD: Measurement using the VOTIS PedCheck system
- PAD patients: Measurement using the VOTIS PedCheck system

SUMMARY:
Feasibility, usability and safety clinical study that is aimed at testing of the non-invasive VOTIS PedCheck system for measurement of changes in absorption of light in order to derive changes in perfusion and oxygen levels in the foot.

DETAILED DESCRIPTION:
Introduction:

Peripheral Arterial Disease (PAD) affects 8-12 million people in the United States, and approximately 230 million worldwide. When linked with diabetes, PAD results in over 71,000 amputations annually.

Patients with PAD have decreased lower extremity arterial perfusion which is commonly referred to as "poor circulation." In most cases of PAD, atherosclerotic plaques narrow the arterial flow lumen which restricts blood flow to the distal extremity. This condition is characterized by progressive vessel obstructions, associated with cardiovascular (CV) events, including myocardial infarction (MI), stroke, limb ischemia, and CV death. Although PAD is a prevalent condition, it is still considered as an underdiagnosed manifestation of atherosclerosis. PAD is one of the most common vascular complications of diabetes, and can cause foot ischemia which is associated with non healing wounds, gangrene and amputations. At present there is no gold standard or test/device to identify, evaluate, and monitor the circulatory health of the foot in a reliable and precise way. In addition, calcification of blood vessels in patients with diabetes complicates the evaluation of perfusion in the foot. Since diabetes has reached epidemic proportions (60M people affected in Europe), there is an urgent need for additional measurement tools for assistance for the evaluation of PAD complications.

The current study is aimed at feasibility, usability and safety testing of the non-invasive VOTIS PedCheck system as an assessment tool of PAD. The protocol allows for 30 PAD patients and 30 self assessed healthy controls.

Objectives:

* To assess the safety of the PedCheck device using HOVR technology
* To calibrate the measurement of changes in absorption of light in order to derive relative perfusion and oxygen levels in the foot.
* To compare between PAD and non-PAD populations using HOVR.

Secondary objective:

• To collect data regarding the usability of the PedCheck device.

Description of investigational product:

Votis PedCheck portable device comprises patches affixed to the foot with encased laser diodes and photodetector sensors that automatically measure absorption of the light. Via lightweight leads, the patches link to a central control and display device. In addition an inflatable blood pressure cuff is placed above the knee. The control device sets the inflation and deflation of the cuff according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Age >40
* Subject must be willing and able to sign an Informed Consent form to participate in the clinical study.

Exclusion Criteria:

* Pregnant and breastfeeding woman
* Any severe concurrent disease which in the judgment of the investigator would make the subject inappropriate for the purposes of this study.

Control group Inclusion Criteria:

• Good health according to self-report

Control group exclusion Criteria:

* History of diabetes and/or a cardiovascular disease according to self-report
* History of heavy smoking (20 cigarettes a day) for at least one year during the last 5 years prior to consent
* Family history of severe cardiovascular disease, i.e. sudden cardiac death below the age of 50, according to self-report
* Use of anti-hypertension drugs

PAD group Inclusion Criteria:

• Subjects who are suspected of having PAD and have undergone or are planned to undergo ABI testing within 60 days prior to or after ICF signature

PAD group exclusion Criteria:

* Existence of a WIfI graded severe foot infection (Infection grade 3) or severe infection (Infection grade 4), i.e. local infection or general infection with signs of systemic inflammatory response syndrome.
* Amputation or a surgical procedure on the foot during the last 2 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be composed of 2 cohorts-
  * Control cohort - Up to 30 healthy non-PAD subjects
  * PAD cohort - Up to 30 PAD patients diagnosed with Peripheral Arterial Disease (PAD)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Severe adverse device effects or serious adverse events that are recorded using standard adverse event report forms | Through study completion, an average of 1 year.
  Observation of adverse skin changes or tissue damage or reports of discomfort.
PedCheck parameters that demonstrate correlation between HOVR and Ankle Brachial Index (ABI) and Toe Brachial Index (TBI). | Through study completion, an average of 1 year.
  HOVR score 0-100. 0-40 being no PAD, 40-100 being increasingly severe PAD.

SECONDARY OUTCOMES:
Evaluation of usability based on collected data using standard convenience scoring questionnaires. | Through study completion, an average of 1 year.
  Usability will be evaluated by standard usability patient and operator questionnaires for scoring convenience. Convenience will be rated by numerical rating scale for scoring convenience 0-5 where 0 represents very hard and 5 very easy.
Evaluation of usability based on collected data using standard pain scoring questionnaires. | Through study completion, an average of 1 year.
  Usability will be evaluated by Numerical rating scale for scoring pain. 0-10 where 0 represents no pain and 10 the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Hamutal Shahar, PhD, Study Director — Votis Subdermal Imaging Technologies
Locations (1):
- Hadassah University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No